CLINICAL TRIAL: NCT04203498
Title: A Double-blind, Randomized, Placebo-controlled, Parallel-group Trial of the Efficacy and Safety of Nabiximols Oromucosal Spray as Add-on Therapy in Patients With Spasticity Due to Multiple Sclerosis
Brief Title: Safety and Effectiveness of Nabiximols Oromucosal Spray as Add-on Therapy in Participants With Spasticity Due to Multiple Sclerosis
Acronym: RELEASE MSS3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated based on a business decision by the Sponsor.
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GWSP18023; 2019-002623-14 (EudraCT Number)
Record Dates: First submitted 2019-12-17; First posted 2019-12-18 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis (MS)
Keywords: Spasticity
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nabiximols (Experimental)
  Interventions: Drug: Nabiximols
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nabiximols — Nabiximols is a complex botanical medicine formulated from extracts of the cannabis plant that contains the principal cannabinoids delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD) and also contains minor constituents, including other cannabinoid and non-cannabinoid plant components, such as terpenes, sterols, and triglycerides.Nabiximols will be self-administered by participants as an oromucosal spray in the morning and evening, up to a maximum of 12 sprays per day for 12 weeks.
  Other Names: GW-1000-02; Sativex
  Arms: Nabiximols
Drug: Placebo — Placebo to match nabiximols will be presented as an oromucosal spray containing the excipients ethanol and propylene glycol (50% v/v) with colorings and flavored with peppermint oil (0.05% v/v). Each spray will deliver 100 microliters (μL) containing no active ingredients. Placebo will be self-administered by participants as an oromucosal spray in the morning and evening, up to a maximum of 12 sprays per day for 12 weeks.
  Arms: Placebo

SUMMARY:
This trial is being conducted to demonstrate the efficacy of nabiximols, compared with placebo, when added to standard of care, in the treatment of muscle spasms associated with multiple sclerosis (MS).

DETAILED DESCRIPTION:
This multicenter, double-blind, placebo-controlled trial includes a 28-day Baseline period, a 12-week treatment period (comprising a 2-week titration phase and a 10-week maintenance phase), and 2-week follow-up period.

Eligible participants will enter the 28-day baseline period. During baseline, participants will maintain their optimized oral MS antispasticity medication regimen and record spasm count using an electronic daily diary. At screening (Day 1), eligible participants will be randomized to either nabiximols or placebo in a 1:1 ratio.

Participants will be advised to titrate the investigational medicinal product (IMP), beginning with 1 spray/day, to an optimized dose or to a maximum of 12 sprays/day over the first 14 days of treatment. Participants may leave a gap between sprays of approximately 15 minutes. Participants should continue at the same dose level achieved at the end of the titration phase ±1 spray divided into a morning dose and an evening dose for the remainder of the treatment period.

Daily spasm count, the participant's symptom experiences, clinician's assessment of spasticity, functional outcomes, health-related quality of life, changes in mood, safety, tolerability, and pharmacokinetics will be evaluated during the treatment period.

Participants who complete the trial will participate for a total of approximately 18 weeks (127 days), including the 28-day baseline period. Participants will have a maximum duration of 85 (±7) days on IMP treatment.

ELIGIBILITY:
Inclusion Criteria:

Criteria at screening:

1. Participant is male or female aged 18 years or above.
2. Participant has had a diagnosis with any disease subtype of multiple sclerosis (MS), by revised 2017 McDonald criteria, for at least 12 months prior to screening and is expected to remain stable for the duration of the trial.
3. Participant has had treatment with at least 1 optimized oral antispasticity therapy prior to Visit 1 that must include either oral baclofen or oral tizanidine (monotherapy or combination therapy).
4. Participant is currently receiving optimized treatment with at least 1 oral antispasticity medication (baclofen, tizanidine, and/or dantrolene) and has been stable for at least 30 days prior to screening.
5. If the participant is currently receiving an approved MS disease-modifying therapy, it must be at a stable dose for at least 3 months prior to screening and is expected to remain stable for the duration of the trial.

Exclusion Criteria:

1. Participant has any concomitant disease or disorder that has spasticity-like symptoms or that may influence the participant's level of spasticity.
2. Participant has had a relapse of MS within the 60 days prior to screening (Visit 1).
3. Participant is currently using or has used cannabis or a cannabinoid-derived product for medicinal or recreational use (within 30 days of screening) and is unwilling to abstain for the duration of the trial.
4. Participant is currently using botulinum toxin injection for the relief of spasticity (within 6 months of screening) and is unwilling to abstain for the duration of the trial.
5. Participant has any known or suspected hypersensitivity to cannabinoids or any of the excipients of the IMP.
6. Participant is male and fertile unless willing to ensure that he uses male contraception or remains sexually abstinent during the trial and for 3 months thereafter.
7. Participant is female and of childbearing potential unless willing to ensure that she uses a highly effective method of birth control during the trial and for 3 months thereafter.
8. Participant is female and pregnant, lactating, or planning pregnancy during the course of the trial or within 3 months thereafter.
9. Participant has received an IMP within the 30 days prior to screening.
10. Participant has a history of severe psychiatric disorder that may be exacerbated by the use of a cannabinoid-containing product.
11. Participant has any known or suspected history of alcohol or substance abuse (including opiate abuse) or dependence within 1 year prior to screening.
12. Participant is currently taking drugs that are solely metabolized by UGT1A9 and UGT2B7.
13. Participant is currently taking strong currently taking strong CYP3A4 inducers (e.g., rifampicin, carbamazepine, phenytoin, phenobarbital, St John's Wort).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (15):
  - University of Alabama at Birmingham School of Medicine, Birmingham, Alabama
  - Neurostudies - Port Charlotte, Port Charlotte, Florida
  - University of South Florida, Tampa, Florida
  - Accel Research Sites - Enterprise, Tampa, Florida
  - Shepherd Center, Atlanta, Georgia
  - Consultants in Neurology - Northbrook, Northbrook, Illinois
  - American Health Network of Indiana, Avon, Indiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - The Multiple Sclerosis Center For Innovations In Care, St Louis, Missouri
  - Raleigh Neurology Associates - Raleigh Location, Raleigh, North Carolina
  - University of Cincinnati (UC) Health, Dayton, Ohio
  - Neurology Clinic - Cordova, Cordova, Tennessee
  - Hope Neurology, Knoxville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
- Czechia (5):
  - Poliklinika Choceň, Choceň, Pardubice
  - Neurologie Taláb Radomír Doc. MUDr., CSc, Hradec Králové
  - Nemocnice Jihlava, Jihlava
  - Fakultní Nemocnice Královské Vinohrady, Prague
  - Krajská Zdravotní - Nemocnice Teplice, Teplice
- Poland (12):
  - Niepubliczny Zakład Opieki Zdrowotnej NEURO - KARD, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne Neuromed - Ośrodek Badań Klinicznych, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Wromedica Centrum Zdrowia, Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne Neuroprotect, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Pratia - Warszawa, Warsaw, Masovian Voivodeship
  - Neuro-Medic Janusz Zbrojkiewicz, Katowice, Silesian Voivodeship
  - Wielospecjalistyczne Centrum Medyczne Ibismed, Zabrze, Silesian Voivodeship
  - SP ZOZ Uniwersytecki Szpital Kliniczny Nr 1 im. Norberta Barlickiego w Łodzi, Lodz
  - Centrum Medyczne Oporów, Lublin
  - Neurologiczny NZOZ Centrum Leczenia SM Ośrodek Badań Klinicznych im. dr n. med. Hanki Hertmanowskiej Witosław Cieślak, Plewiska
  - Wromedica Centrum Zdrowia, Wroclaw
  - RESMEDICA Poradnia Neurologiczna, Kielce, Świętokrzyskie Voivodeship
- Romania (4):
  - Centrul Medical Clubul Sanatatii, Campulung Muscel
  - Spitalul Municipal Caracal, Caracal
  - Spitalul Clinic Cai Ferate Constanta, Constanța
  - Spitalul Municipal Sf. Dr. Cosma si Damian Radauti, Radauti
- Barts Health NHS Trust, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nabiximols: Patients randomized to receive GW-1000-2 (nabiximols) self-administered as an oromucosal spray in the morning and evening, up to a maximum of 12 sprays per day for 12 weeks.
- Placebo: Patients randomized to receive placebo self-administered as an oromucosal spray in the morning and evening, up to a maximum of 12 sprays per day for 12 weeks.
Period: Overall Study
Arm/Group | Nabiximols | Placebo
Started | 69 | 70
Safety Analysis Set | 67 | 70
Completed | 55 | 66
Not Completed | 14 | 4
Not completed — Decision by the investigator, GW, or authority | 0 | 1
Not completed — Withdrawal of patient consent | 7 | 2
Not completed — Adverse Event | 4 | 1
Not completed — Drug not dispensed due to endpoint error | 1 | 0
Not completed — Did not receive IMP | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported from the Full Analysis Set defined as all patients from the Safety Analysis Set who signed the informed consent and are randomized by interactive response technology.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nabiximols | Placebo | Total
Number analyzed (Participants) | 67 | 70 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (10.4) | 53.0 (10.2) | 52.6 (10.2)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0
  ≥18 years to <45 years | 14 | 15 | 29
  ≥45 years to <65 years | 44 | 46 | 90
  ≥65 years | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 52 | 95
  Male | 24 | 18 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 62 | 68 | 130
  Black or African American | 3 | 1 | 4
  Asian | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Daily Spasm Count From Baseline to Week 12 By 4-Week Period During the 12-Week Randomized Period
Description: The change in the average daily spasm count was assessed compared to the baseline period.
Time Frame: Baseline to Week 12
Population: Average daily spasm count was assessed in participants with available data in the Full Analysis Set defined as all patients from the Safety Analysis Set who signed the informed consent and are randomized by interactive response technology..
Measure: Least Squares Mean (Standard Error); unit: daily spasm count
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 67 | 70
daily spasm count
  Week 1 to 4 | -2.23 (0.412) | -1.62 (0.394)
  Week 5 to 8: number analyzed (Participants) | 59 | 67
  Week 5 to 8 | -3.42 (0.607) | -2.62 (0.583)
  Week 9 to 12: number analyzed (Participants) | 55 | 65
  Week 9 to 12 | -3.84 (0.689) | -3.11 (0.659)
Statistical Analysis 1: Comparison: Nabiximols vs Placebo; Week 9 to 12 (primary outcome statistics); Test type: Superiority; p = 0.4263, Linear mixed model repeated measures; Difference in least squares means = -0.73, 95% CI 2-sided [-2.54 to 1.08], Standard Error of Mean 0.914

2. Secondary Outcome: Change in Multiple Sclerosis Spasticity Scale (MSSS-88) Total Score
Description: The MSSS-88 is a self-reported measure of the impact of spasticity (muscle stiffness and spasms) in MS. This 88-item scale captures the patient experience and impact of spasticity, including muscle stiffness, pain and discomfort, muscle spasms, effect on daily activities, ability to walk, body movement, patient feelings, and social functioning. Responses to individual questions can range from "1 - not at all bothered" to "4 - extremely bothered", ranging from 88 to 352 total score. Scores are summed and higher scores indicate poor clinical outcome. Least square means are being reported, with greater negative values indicating better outcome.
Time Frame: Week 8 and Week 12
Population: Changes in Multiple Sclerosis Spasticity Scale were assessed in participants with available data in the Full Analysis Set defined as all patients from the Safety Analysis Set who signed the informed consent and are randomized by interactive response technology.
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 51 | 54
unit on a scale
  Week 8 | -21.64 (5.775) | -26.11 (5.461)
  Week 12: number analyzed (Participants) | 46 | 51
  Week 12 | -26.53 (5.807) | -23.18 (5.426)

3. Secondary Outcome: Number of Patients Reporting Any Treatment-emergent Adverse Events
Description: A TEAE is an adverse event that started, or worsened in severity or seriousness, following the first dose of the investigational medicinal product.
Time Frame: From date of first dose of IMP up to 30 days after last dose, up to approximately 16 weeks
Population: Treatment-emergent adverse events were assessed in the Safety Analysis Set defined as all participants who received at least 1 dose of study intervention in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 67 | 70
Participants | 47 | 32

4. Secondary Outcome: Change From Baseline in Clinical Laboratory Test Values
Time Frame: Baseline up to Week 12
Population: Clinical laboratory values were assessed in patients with available data in the Safety Analysis Set defined as all participants who received at least 1 dose of study intervention in the study.
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 59 | 62
10^9 cells/liter
  Basophils | -0.009 (0.030) | 0.002 (0.037)
  Eosinophils | -0.007 (0.110) | 0.006 (0.086)
  Leukocytes | 0.146 (1.095) | 0.139 (1.881)
  Lymphocytes | -0.056 (0.368) | 0.009 (0.315)
  Monocytes | 0 (0.120) | 0.001 (0.126)
  Neutrophils | 0.217 (1.004) | 0.083 (1.788)
  Platelets | -0.085 (42.392) | 5.290 (49.972)

5. Secondary Outcome: Change From Baseline in Erythrocytes
Time Frame: Baseline up to Week 12
Population: Erythrocytes were assessed in patients with available data in the Safety Analysis Set defined as all participants who received at least 1 dose of study intervention in the study.
Measure: Mean (Standard Deviation); unit: 10^12 cells/liter
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 59 | 62
10^12 cells/liter | 0.010 (0.241) | -0.007 (0.251)

6. Secondary Outcome: Change From Baseline in Hemoglobin
Time Frame: Baseline up to Week 12
Population: Hemoglobin was assessed in patients with available data in the Safety Analysis Set defined as all participants who received at least 1 dose of study intervention in the study.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 59 | 62
g/dL | -0.025 (0.735) | -0.021 (0.726)

7. Secondary Outcome: Change From Baseline in Hematocrit Ratio
Description: The hematocrit ratio measures the volume of red blood cells compared to the total blood volume.
Time Frame: Baseline up to Week 12
Population: Hematocrit ratio was assessed in patients with available data in the Safety Analysis Set defined as all participants who received at least 1 dose of study intervention in the study.
Measure: Mean (Standard Deviation); unit: ratio of packed cells to total volume
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 59 | 62
ratio of packed cells to total volume | -0.002 (0.025) | -0.002 (0.027)

8. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Hemoglobin
Time Frame: Baseline up to Week 12
Population: Erythrocyte mean corpuscular hemoglobin was assessed patients with available data in the Safety Analysis Set defined as all participants who received at least 1 dose of study intervention in the study.
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 59 | 62
pg | -0.156 (0.608) | -0.005 (0.881)

9. Secondary Outcome: Change From Baseline in Blood Pressure
Time Frame: Baseline up to Week 12
Population: Blood pressure was assessed in patients with available data in the Safety Analysis Set defined as all participants who received at least 1 dose of study intervention in the study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 60 | 67
mmHg
  Systolic Blood Pressure | -1.6 (10.95) | 2.6 (11.31)
  Diastolic Blood Pressure | 0.3 (8.20) | 2.7 (13.38)

10. Secondary Outcome: Change From Baseline in Heart Rate
Time Frame: Baseline up to Week 12
Population: Heart rate was assessed in patients with available data in the Safety Analysis Set defined as all participants who received at least 1 dose of study intervention in the study.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 60 | 67
beats/minute | 2.5 (7.70) | 0.4 (10.14)

11. Secondary Outcome: Change From Baseline in Electrocardiogram Parameters
Time Frame: Baseline up to Week 12
Population: Electrocardiogram parameters were assessed in patients with available data in the Safety Analysis Set. defined as all participants who received at least 1 dose of study intervention in the study.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 61 | 67
msec
  PR interval, aggregate | 5.5 (20.51) | 1.3 (21.05)
  QRS duration | 1.9 (9.89) | -6.5 (37.08)
  QTcB interval: number analyzed (Participants) | 60 | 66
  QTcB interval | 1.5 (29.58) | -2.4 (33.29)
  QTcF interval: number analyzed (Participants) | 60 | 67
  QTcF interval | 2.9 (26.69) | -3.2 (32.40)

12. Secondary Outcome: Change From Baseline in Electrocardiogram Pulse Rate
Time Frame: Baseline up to Week 12
Population: Electrocardiogram heart rate was assessed in patients with available data in the Safety Analysis Set defined as all participants who received at least 1 dose of study intervention in the study.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 61 | 67
beats/min | -2.6 (10.21) | 0.5 (8.74)

13. Secondary Outcome: Change From Baseline in Weight
Time Frame: Baseline up to Week 12
Population: Weight was assessed in patients with available data in the Safety Analysis Set defined as all participants who received at least 1 dose of study intervention in the study.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 59 | 67
kg | -0.338 (3.198) | -0.394 (3.578)

14. Secondary Outcome: Change in Body Mass Index
Time Frame: Baseline up to Week 12
Population: Body mass index was assessed in patients with available data in the Safety Analysis Set defined as all participants who received at least 1 dose of study intervention in the study.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 59 | 67
kg/m^2 | -0.086 (1.052) | -0.159 (1.287)

15. Secondary Outcome: Number of Patients With Suicidal Ideation or Behavior Based on Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a short questionnaire that is used to assess suicidal ideation (5 questions) and behavior (5 questions) since last patient visit. The questionnaire is completed by participants answering yes or no to each question.
Time Frame: Screening up to Week 12
Population: Suicidal ideation or behavior was assessed in the Safety Analysis Set. defined as all participants who received at least 1 dose of study intervention in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Nabiximols | Placebo
Number analyzed (Participants) | 67 | 70
Participants
  Screening: Ideation, Wish to be dead | 1 | 1
  Screening: Ideation, Non-specific active thoughts | 1 | 1
  Screening: Ideation, Active any method no intent | 0 | 1
  Screening: Ideation, Active intent to act, no plan | 0 | 0
  Screening: Ideation, Active specific plan/intent | 0 | 0
  Screening: Behavior, Preparatory acts or behavior | 0 | 0
  Screening: Behavior, Aborted attempt | 0 | 0
  Screening: Behavior, Interrupted attempt | 0 | 0
  Screening: Behavior, Actual attempt | 0 | 1
  Screening: Behavior, Completed suicide | 0 | 0
  Screening: Suicidal ideation or behavior | 1 | 1
  Screening: Self-injurious behavior without suicidal intent | 0 | 0
  Baseline: Ideation, Wish to be dead | 0 | 0
  Baseline: Ideation, Non-specific active thoughts | 0 | 0
  Baseline: Ideation, Active any method no intent | 0 | 0
  Baseline: Ideation, Active intent to act, no plan | 0 | 0
  Baseline: Ideation, Active specific plan/intent | 0 | 0
  Baseline: Behavior, Preparatory acts or behavior | 0 | 0
  Baseline: Behavior, Aborted attempt | 0 | 0
  Baseline: Behavior, Interrupted attempt | 0 | 0
  Baseline: Behavior, Actual attempt | 0 | 0
  Baseline: Behavior, Completed suicide | 0 | 0
  Baseline: Suicidal ideation or behavior | 0 | 0
  Baseline: Self-injurious behavior without suicidal intent | 0 | 0
  Week 2: Ideation, Wish to be dead | 1 | 0
  Week 2: Ideation, Non-specific active thoughts | 0 | 0
  Week 2: Ideation, Active any method no intent | 0 | 0
  Week 2: Ideation, Active intent to act, no plan | 0 | 0
  Week 2: Ideation, Active specific plan/intent | 0 | 0
  Week 2: Behavior, Preparatory acts or behavior | 0 | 0
  Week 2: Behavior, Aborted attempt | 0 | 0
  Week 2: Behavior, Interrupted attempt | 0 | 0
  Week 2: Behavior, Actual attempt | 0 | 0
  Week 2: Behavior, Completed suicide | 0 | 0
  Week 2: Suicidal ideation or behavior | 1 | 0
  Week 2: Self-injurious behavior without suicidal intent | 0 | 0
  Week 4: Ideation, Wish to be dead | 0 | 0
  Week 4: Ideation, Non-specific active thoughts | 0 | 0
  Week 4: Ideation, Active any method no intent | 0 | 0
  Week 4: Ideation, Active intent to act, no plan | 0 | 0
  Week 4: Ideation, Active specific plan/intent | 0 | 0
  Week 4: Behavior, Preparatory acts or behavior | 0 | 0
  Week 4: Behavior, Aborted attempt | 0 | 0
  Week 4: Behavior, Interrupted attempt | 0 | 0
  Week 4: Behavior, Actual attempt | 0 | 0
  Week 4: Behavior, Completed suicide | 0 | 0
  Week 4: Suicidal ideation or behavior | 0 | 0
  Week 4: Self-injurious behavior without suicidal intent | 0 | 0
  Week 8: Ideation, Wish to be dead | 0 | 0
  Week 8: Ideation, Non-specific active thoughts | 0 | 0
  Week 8: Ideation, Active any method no intent | 0 | 0
  Week 8: Ideation, Active intent to act, no plan | 0 | 0
  Week 8: Ideation, Active specific plan/intent | 0 | 0
  Week 8: Behavior, Preparatory acts or behavior | 0 | 0
  Week 8: Behavior, Aborted attempt | 0 | 0
  Week 8: Behavior, Interrupted attempt | 0 | 0
  Week 8: Behavior, Actual attempt | 0 | 0
  Week 8: Behavior, Completed suicide | 0 | 0
  Week 8: Suicidal ideation or behavior | 0 | 0
  Week 8: Self-injurious behavior without suicidal intent | 0 | 0
  Week 12: Ideation, Wish to be dead | 0 | 0
  Week 12: Ideation, Non-specific active thoughts | 0 | 0
  Week 12: Ideation, Active any method no intent | 0 | 0
  Week 12: Ideation, Active intent to act, no plan | 0 | 0
  Week 12: Ideation, Active specific plan/intent | 0 | 0
  Week 12: Behavior, Preparatory acts or behavior | 0 | 0
  Week 12: Behavior, Aborted attempt | 0 | 0
  Week 12: Behavior, Interrupted attempt | 0 | 0
  Week 12: Behavior, Actual attempt | 0 | 0
  Week 12: Behavior, Completed suicide | 0 | 0
  Week 12: Suicidal ideation or behavior | 0 | 0
  Week 12: Self-injurious behavior without suicidal intent | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline up to 14 days after the end of treatment visit, up to Day 99 (safety follow up visit).
Arm/Group | Nabiximols | Placebo
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/70
Serious Adverse Events (participants affected / at risk) | 3/67 | 5/70
Other Adverse Events (participants affected / at risk) | 46/67 | 19/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nabiximols (N=67) | Placebo (N=70)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nabiximols (N=67) | Placebo (N=70)
Dizziness (Nervous system disorders) | 14 (15) | 5 (8)
Fatigue (General disorders) | 8 (9) | 2 (3)
Somnolence (Nervous system disorders) | 7 (7) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 6 (8) | 0 (0)
Asthenia (General disorders) | 4 (4) | 2 (2)
Taste disorder (Nervous system disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (5)
Urinary tract infection (Infections and infestations) | 3 (3) | 4 (5)

LIMITATIONS AND CAVEATS:
Study enrollment was ended early and did not reach the planned number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT04203498/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT04203498/SAP_001.pdf